CLINICAL TRIAL: NCT03732495
Title: A Prospective, Multicentre Phase II Study of the Efficacy of Lenvatinib Combined With Denosumab in the Treatment of Patients With Predominant Bone Metastatic Radioiodine Refractory Differentiated Thyroid Carcinomas (LENVOS)
Brief Title: Study of the Efficacy of Lenvatinib Combined With Denosumab in the Treatment of Patients With Predominant Bone Metastatic Radioiodine Refractory Differentiated Thyroid Carcinomas
Acronym: LENVOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET17-191
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Cancer Metastatic
MeSH Terms: interventions — lenvatinib; Denosumab

STUDY DESIGN:
Intervention Model Description: Patients with predominant bone metastases from Radioiodine-Refractory Differentiated Thyroid Carcinoma (RR-DTC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial arm (Experimental): Lenvatinib and Denosumab will be used in the indication of their respective SmPCs.
  Study treatments will be divided in fictitious cycles of 28 days. Lenvatinib and Denosumab will be administered as per investigator's decision, based on the data from their SmPC, at starting doses of 24mg once daily and 120mg once every 4 weeks, respectively. Dose modification guidelines of their respective SmPCs will apply.
  Lenvatinib should be started the day after the inclusion. It will be taken every day at the same time, preferentially in the morning.
  As in routine practice, all patients will be supplemented with daily doses of at least 500mg Calcium and 400IU Vitamin D, unless hypercalcemia is present.
  Patients will be encouraged to maintain good oral hygiene during treatment with Denosumab.
  Study drugs will be continued until a treatment discontinuation criterion is met.
  Interventions: Drug: Lenvatinib + Denosumab

INTERVENTIONS:
Drug: Lenvatinib + Denosumab — Lenvatinib and Denosumab will be used in the indication of their respective SmPCs.
  Study treatments will be divided in fictitious cycles of 28 days. Lenvatinib and Denosumab will be administered as per investigator's decision, based on the data from their SmPC, at starting doses of 24mg once daily and 120mg once every 4 weeks, respectively. Dose modification guidelines of their respective SmPCs will apply.
  Lenvatinib should be started the day after the inclusion. It will be taken every day at the same time, preferentially in the morning.
  As in routine practice, all patients will be supplemented with daily doses of at least 500mg Calcium and 400IU Vitamin D, unless hypercalcemia is present.
  Patients will be encouraged to maintain good oral hygiene during treatment with Denosumab.
  Study drugs will be continued until a treatment discontinuation criterion is met

SUMMARY:
This study evaluates the combination of lenvatinib with denosumab in bone-predominant metastatic Radioiodine Refractory Differentiated Thyroid Carcinomas. All patients will receive this combination of treatments.

DETAILED DESCRIPTION:
Patients are usually considered for directed therapy (radiotherapy and/or surgery and/or thermo-ablation) in case of symptomatic lesions or at high risk of local complications. They also usually receive systemic bone-directed agents (bisphosphonate or denosumab), despite sparse available data in the context of differentiated thyroid carcinomas (DTC). As bone-directed agents have no antitumor activity, patients may require additional treatments. To date, only sorafenib and lenvatinib have been approved in the treatment of advanced Radioiodine Refractory Differentiated Thyroid Carcinomas (RR-DTC).

Lenvatinib demonstrated efficacy in RR-DTC compared to placebo. While other kinase inhibitors appeared to be less effective in controlling bone metastatic disease compared to other soft tissue sites, lenvatinib showed, in a small number of patients, significant decrease in bone tumors size.

Even if both study drugs are indicated in the treatment of patients suffering from RR-DTC with bone metastases, it is of essential importance to confirm that lenvatinib can provide clinical benefit and antitumor activity when combined with denosumab in this population.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of 18 years of age or older at the day of consenting to the study;
* I2. Patients with follicular cell-derived thyroid (papillary, vesicular or and poorly differentiated);
* Radioiodine-Refractory disease as defined by at least one of the following :

  * Presence of malignant/metastatic tissue that does not concentrate radioiodine (RAI),
  * Loss by the tumor tissue of the ability to concentrate RAI after previous evidence of RAI-avid disease,
  * Concentration of RAI in some lesions but not in others,
  * Progression of metastatic disease despite significant concentration of RAI;
* Predominant bone metastases (without threatening extra-bone metastasis)
* Patient at risk of Skeletal-Related Event defined by the occurrence of at least one of the following event within 12 months prior to inclusion:

  * Skeletal-Related Event, including indication of loco regional procedure (i.e. radiation therapy, interventional radiology),
  * Progressive disease with measurable metastatic bone lesion(s) as per the RECIST1.1; Nota Bene: bone lesions with soft tissue involvement are considered as measurable.
* Performance Status of the Eastern Cooperative Oncology Group (ECOG) ≤2;
* Adequate organ function within 14 days prior to treatment start, defined as the following:

  * Neutrophils count ≥ 1.5 Gi/l
  * Hemoglobin ≥ 9.0 g/dl
  * Platelets count ≥ 100 Gi/l
  * Prothrombin Time (PT) ≤ 1.2 x ULN or International Normalized Ratio ≤ 1.5 Nota bene: Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the targeted anticoagulation.
  * Serum transaminases (ASAT and ALAT) ≤ 3.0 x upper limit of the normal (ULN) (5.0 x ULN in case of liver metastases)
  * Serum total bilirubin ≤ 2 x ULN
  * Creatinine clearance ≥ 30ml/min;
  * Absence of proteinuria Nota Bene: patients with proteinuria ≥1+ on dipstick urinalysis will have to undergo 24 hours urine collection. Subjects with urine protein ≥1g/24h will be ineligible;
  * Albumin-adjusted serum calcium ≥ 2.0 mmol/l (8.0mg/dl) and ≤ 2.9 mmol/l (11.5mg/dl)
* Patient and his/her partner using 2 forms of effective contraception:

  * For women of child-bearing potential: at least 4 weeks prior to study entry, during the study participation and for at least 1 month post-lenvatinib and at least 5 months post-denosumab,
  * For men: at least 4 weeks prior to study entry and during the study participation;
* Patient must be covered by a medical insurance;
* Willingness and ability to comply with the study requirements;
* Signed and dated informed consent indicating that the patient has been informed of all the aspects of the trial prior to enrolment.

Non-inclusion Criteria:

* Histological diagnosis of the following DTC subtypes: medullar, anaplastic, lymphoma or sarcoma;
* Prior history of malignancies other than study disease within the last 3 years, except locally curable disease with no sign of relapse;
* Prior or current treatment with denosumab or any other bone-directed agent (including bisphosphonates), regardless of the indication;
* Prior or current treatment with any tyrosine kinase inhibitor, including but not limited to lenvatinib and denosumab ;
* Patient with imminent or confirmed Skeletal-Related Event as defined in the protocol;
* Uncontrolled arterial hypertension (150mmHg/90mmHg) despite an optimal antihypertensive intervention; patients with high blood pressure can be enrolled provided that the hypertension is well controlled at a stable dose of antihypertensive therapy for at least 1 week prior to lenvatinib start;
* Any condition leading to an increased risk of bleeding or hemorrhage;
* Any other contraindication to lenvatinib and/or denosumab
* Major surgery within 3 weeks prior to the first study drug administration or major surgery planned during the course of the study;
* Unhealed lesion from dental or oral surgery;
* Any dental or jaw condition that may lead or already led to osteonecrosis of the jaw or to oral surgery; Nota Bene: a consultation with a specialist must confirm that dental and oral cavity assessment allows starting a treatment with denosumab.
* Any active infection, including known infection with HIV, Hepatitis B or Hepatitis C;
* Patient participating to a clinical trial that can interfere with the primary outcome assessment or treatment with any investigational drug within 4 weeks prior to the start date of study drugs or planned during the study participation;
* Any organic or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results;
* Pregnant or breast feeding women. Women of childbearing potential* are required to have a negative serum pregnancy test within 72 hours prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test

  *: Female patients who meet at least one of the following criteria are defined as women of non-childbearing potential:
  * ≥50 years old and naturally amenorrheic for ≥ 1 year
  * Permanent premature ovarian failure confirmed by a specialist gynecologist
  * Previous bilateral salpingo-oophrectomy
  * XY genotype, Turner's syndrome, or uterine agenesis Female patients who do not meet at least one of the above criteria are defined as women of childbearing potential.
* Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of lenvatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection);
* Patient with history or active gastrointestinal or non-gastrointestinal fistula;
* Hypersensitivity or history of allergic reactions attributed to compounds of similar chemical or biologic composition of study drugs ;
* History or active significant cardiovascular impairment : congestive heart failure greater than New York Heart Association class II, unstable angina, myocardial infarction, stroke, or cardiac arrhythmia associated with impairment within 6 months of the first dose of study drug;
* Clinically significant electrocardiogram abnormality, including marked baseline prolonged QT/QTc interval (e.g., a repeated demonstration of a QTc interval > 500 msec);
* Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results.
* Patients using prohibited concomitant and/or concurrent medications.
* Patient requiring tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Determination of the efficacy of lenvatinib associated with denosumab in the treatment of patients with predominant bone metastases from Radioiodine-Refractory Differentiated Thyroid Carcinoma | 24 months
  The 24-month Skeletal-Related Event-Free (24M-SREF) rate will be defined as the proportion of patients without occurrence of new bone metastatic lesions at 24 months
Determination of the efficacy of lenvatinib associated with denosumab in the treatment of patients with predominant bone metastases from Radioiodine-Refractory Differentiated Thyroid Carcinoma | 24 months
  The 24-month Skeletal-Related Event-Free (24M-SREF) rate will be defined as the proportion of patients without pathological bone fracture (either vertebral or non-vertebral) at 24 months
Determination of the efficacy of lenvatinib associated with denosumab in the treatment of patients with predominant bone metastases from Radioiodine-Refractory Differentiated Thyroid Carcinoma | 24 months
  The 24-month Skeletal-Related Event-Free (24M-SREF) rate will be defined as the proportion of patients without spinal cord compression at 24 months
Determination of the efficacy of lenvatinib associated with denosumab in the treatment of patients with predominant bone metastases from Radioiodine-Refractory Differentiated Thyroid Carcinoma | 24 months
  The 24-month Skeletal-Related Event-Free (24M-SREF) rate will be defined as the proportion of patients without bone-related orthopedic surgical intervention at 24 months

SECONDARY OUTCOMES:
Determination of the progression free survival | 24 months
  Progression-Free Survival will be defined as the time from the date of inclusion to the date of first documented progression or death due to any cause
Determination of the objective response rate | 24 months
  Objective Response Rate will be defined as the proportion of patients with a best overall response of Complete Response or Partial Response during the study
Determination of the time to the first local procedure | 24 months
  Time to the first local procedure will be defined as the time from the date of inclusion to the date of any local procedure (external beam radiation therapy, thermoablation, cementoplasty…) aiming at relieving bone-related symptoms
Determination of the time to treatment failure | 24 months
  Time to Treatment Failure will be measured from the time of inclusion until discontinuation of treatment for any reason other than 'protocol deviation' or 'administrative problems', including SRE, clinical deterioration, treatment toxicity, and death.
Determination of the analgesic consumption | 24 months
  Analgesic consumption will be assessed and presented in morphine equivalent by 24 hours
Determination of the Quality of life using European Organisation for Research and Treatment of Cancer (EORTC) questionnaire | 24 months
  Using the EORTC QLQ-C30 (Quality of Life Questionnaire) - Scale range: 1 (better outcome) to 4 (worse outcome) for 28 variables and from 1 (better outcome) to 7 (worse outcome) for 2 variables
Determination of the Quality of life using European Organisation for Research and Treatment of Cancer (EORTC) questionnaire | 24 months
  Using the EORTC QLQ-BM22 (Bone Metastasis module) - Scale range 1 (better outcome) to 4 (worse outcome) for 22 items.
Determination of the tolerance profile | 24 months
  Tolerance profile will be described through the incidence and severity of drug-related adverse events (AE), AESI, SAE and deaths according to the last version of the NCI-CTC AE classification

OTHER OUTCOMES:
Determination of predictive biomarker of tumor response | 24 months
  Serum levels of Carboxy-terminal collagen crosslinks
Determination of predictive biomarker of tumor response | 24 months
  Serum levels of osteocalcin
Determination of predictive biomarker of tumor response | 24 months
  Serum levels of bone alkaline phosphatases
Determination of predictive biomarker of tumor response | 24 months
  Serum levels of osteoprotegerin
Determination of predictive biomarker of tumor response | 24 months
  Serum levels of soluble receptor activator of nuclear factor-kB ligand
Determination of predictive factors of tumor response | 14 days
  Levels of tumor perfusion (ml/minute) associated with anti-tumor efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Christelle De La Fouchardiere, MD, Principal Investigator — Centre Leon Berard
Locations (14):
- France (14):
  - CHU Angers, Angers
  - CHRU Besançon, Besançon
  - CHU Bordeaux - Hôpital Saint-André, Bordeaux
  - Institut Bergonie, Bordeaux
  - Hospices Civils de Lyon - Groupement Hospitalier Est, Bron
  - Centre Geogres François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - APHP Saint Louis, Paris
  - APHP La Pitié Salpétrière, Paris
  - Institut Jean Godinot, Reims
  - Institut du Cancer Strasbourg (ICANS), Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif